CLINICAL TRIAL: NCT02808923
Title: Effects of Long-term Foam Rolling Compared to Static Stretching on Hamstring Muscle Flexibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 908292-1
Record Dates: First submitted 2016-06-15; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Muscle Hypertonia
MeSH Terms: conditions — Muscle Hypertonia | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Foam rolling (Experimental): Participants in the foam rolling group will perform unilateral rolling of the hamstring musculature from ischial tuberosity to posterior knee in supine for 2 repetitions of 1 minute with 15 second rest between repetitions at a consistent cadence of 1 second superiorly and 1 second inferiorly. Subjects will be asked to adjust pressure as needed to maintain a consistent moderate pressure on the treatment area. Participants will use new and individually issued high density foam rollers that are 6" diameter x 36" length.
  Interventions: Other: Foam Rolling
- Static stretching (Experimental): Participants in the static stretching group will perform sustained static hamstring stretching for 2 repetitions of 1 minute bouts for the same leg before switching sides using moderate pressure in supine against the wall. Subjects will rest for 15 seconds between repetitions and adjust distance from the wall to perceive moderate intensity.
  Interventions: Other: Static Stretching
- Control (No Intervention): The control group will perform their regular baseline activities without the addition of a specific lower extremity flexibility program. If the subjects are currently performing stretching of any mode at baseline, they will be allowed to continue with that activity.

INTERVENTIONS:
Other: Foam Rolling — Participants will perform unilateral hamstring rolling for 2 repetitions of 1 minute with 15 second rest breaks on each leg with a 6"x 36" foam roller.
  Arms: Foam rolling
Other: Static Stretching — Participants will perform supine static hamstring stretch on a wall for 2 repetitions of 1 minute with 15 second rest breaks on each leg. When the position no longer causes a moderate stretching sensation to the hamstring, subjects will move their bodies closer to the wall to intensify the stretch.
  Arms: Static stretching

SUMMARY:
The purpose of this study to to compare the long-term effects of foam rolling in comparison to static stretching and a control group on hamstring flexibility. The investigators hypothesize that participants in the foam rolling and static stretching group will demonstrate increased flexibility to the control group, but will a difference will not be observed between the foam rolling and static stretching groups.

ELIGIBILITY:
Inclusion Criteria:

* Active 90/90 hamstring length goniometric measurement of greater than 10 degrees at baseline
* Active straight leg raise of less than 90 degrees

Exclusion Criteria:

* History of lower extremity injury including but not limited to sprain, strain, fracture, or any surgical intervention that lead to a decrease in activity greater than two weeks within the last six months
* Current involvement in a lower extremity flexibility program outside of their regular activity

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in 90/90 hamstring length | Baseline, 3 weeks, 6 weeks
  Participant is supine, hip flexed to 90 degrees, knee extension range of motion measured actively from 90 degree starting position with a standard goniometer

SECONDARY OUTCOMES:
Change in Active straight leg raise - Range of motion | Baseline, 3 weeks, 6 weeks
  Participant is supine, with contralateral leg straight the participant will actively raise the leg until end of range with hip flexion being measured by goniometer
Change in Active straight leg raise - Functional Movement Screen | Baseline, 3 weeks, 6 weeks
  Participant is supine, with contralateral leg straight the participant will actively raise the leg until end of range. This end range will be compared to a standardized position using a dowel and will be scored according to the functional movement screen.
Change in Sit-and-reach | Baseline, 3 weeks, 6 weeks
  Using a standardized sit-and-reach box, participants will sit with legs together, knees extended, and hands overlapped and extended in front of the body. The subject will forward flex until end range of motion measured in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Schongalla, DPT, Principal Investigator — Creighton University

IPD SHARING:
Plan to Share IPD: Yes
Non-identifying participant demographics and data on outcome measures (range of motion) for the study may be made available through publication or presentation on the study.

REFERENCES:
- [Background] Mistry GS, Vyas NJ, Sheth, MS. Comparison of hamstrings flexibility in subjects with chronic low back pain versus normal individuals. J Clin Exp Res. 2014; 2(1): 85-88.
- [Background] Barnes. The Basic Science Myofascial Release: Morphologic Change in Connective Tissue. Journal of Bodywork and Movement Therapies. 1997;1(4):231-238.
- [Background] Cunha AC, Burke TN, Franca FJ, Marques AP. Effect of global posture reeducation and of static stretching on pain, range of motion, and quality of life in women with chronic neck pain: a randomized clinical trial. Clinics (Sao Paulo). 2008 Dec;63(6):763-70. doi: 10.1590/s1807-59322008000600010. PMID 19060998
- [Background] Cheatham SW, Kolber MJ, Cain M, Lee M. THE EFFECTS OF SELF-MYOFASCIAL RELEASE USING A FOAM ROLL OR ROLLER MASSAGER ON JOINT RANGE OF MOTION, MUSCLE RECOVERY, AND PERFORMANCE: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2015 Nov;10(6):827-38. PMID 26618062
- [Background] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684
- [Background] Chan SP, Hong Y, Robinson PD. Flexibility and passive resistance of the hamstrings of young adults using two different static stretching protocols. Scand J Med Sci Sports. 2001 Apr;11(2):81-6. doi: 10.1034/j.1600-0838.2001.011002081.x. PMID 11252465
- [Background] Schleip R. Fascial plasticity - a new neurobiological explanation: Part 1. Jounral of Bodywork and Movement Therapies. 2003;7(1): 11-19.
- [Background] MacDonald GZ, Penney MD, Mullaley ME, Cuconato AL, Drake CD, Behm DG, Button DC. An acute bout of self-myofascial release increases range of motion without a subsequent decrease in muscle activation or force. J Strength Cond Res. 2013 Mar;27(3):812-21. doi: 10.1519/JSC.0b013e31825c2bc1. PMID 22580977
- [Background] Sullivan KM, Silvey DB, Button DC, Behm DG. Roller-massager application to the hamstrings increases sit-and-reach range of motion within five to ten seconds without performance impairments. Int J Sports Phys Ther. 2013 Jun;8(3):228-36. PMID 23772339
- [Background] Pearcey GE, Bradbury-Squires DJ, Kawamoto JE, Drinkwater EJ, Behm DG, Button DC. Foam rolling for delayed-onset muscle soreness and recovery of dynamic performance measures. J Athl Train. 2015 Jan;50(1):5-13. doi: 10.4085/1062-6050-50.1.01. Epub 2014 Nov 21. PMID 25415413
- [Background] Skarabot J, Beardsley C, Stirn I. Comparing the effects of self-myofascial release with static stretching on ankle range-of-motion in adolescent athletes. Int J Sports Phys Ther. 2015 Apr;10(2):203-12. PMID 25883869
- [Background] Peacock CA, Krein DD, Antonio J, Sanders GJ, Silver TA, Colas M. Comparing Acute Bouts of Sagittal Plane Progression Foam Rolling vs. Frontal Plane Progression Foam Rolling. J Strength Cond Res. 2015 Aug;29(8):2310-5. doi: 10.1519/JSC.0000000000000867. PMID 25647651
- [Background] Healey KC, Hatfield DL, Blanpied P, Dorfman LR, Riebe D. The effects of myofascial release with foam rolling on performance. J Strength Cond Res. 2014 Jan;28(1):61-8. doi: 10.1519/JSC.0b013e3182956569. PMID 23588488
- [Background] Halperin I, Aboodarda SJ, Button DC, Andersen LL, Behm DG. Roller massager improves range of motion of plantar flexor muscles without subsequent decreases in force parameters. Int J Sports Phys Ther. 2014 Feb;9(1):92-102. PMID 24567860
- [Background] Junker DH, Stoggl TL. The Foam Roll as a Tool to Improve Hamstring Flexibility. J Strength Cond Res. 2015 Dec;29(12):3480-5. doi: 10.1519/JSC.0000000000001007. PMID 25992660
- [Background] Miller MK, Ashley RM. Foam Rollers Show No Increase in the Flexibility of the Hamstring Muscle Group. Journal of Undergraduate Research. 2006; 10: 1-4.
- [Background] Goldspink G. Cellular and molecular aspects of adaptation in skeletal muscle. In: Komi PV, editor. Strength and Power in Sports. Oxford: Blackwell, 1992:211-29.
- [Background] Magnusson SP, Simonsen EB, Aagaard P, Sorensen H, Kjaer M. A mechanism for altered flexibility in human skeletal muscle. J Physiol. 1996 Nov 15;497 ( Pt 1)(Pt 1):291-8. doi: 10.1113/jphysiol.1996.sp021768. PMID 8951730
- [Background] Jay K, Sundstrup E, Sondergaard SD, Behm D, Brandt M, Saervoll CA, Jakobsen MD, Andersen LL. Specific and cross over effects of massage for muscle soreness: randomized controlled trial. Int J Sports Phys Ther. 2014 Feb;9(1):82-91. PMID 24567859
- [Background] Law RY, Harvey LA, Nicholas MK, Tonkin L, De Sousa M, Finniss DG. Stretch exercises increase tolerance to stretch in patients with chronic musculoskeletal pain: a randomized controlled trial. Phys Ther. 2009 Oct;89(10):1016-26. doi: 10.2522/ptj.20090056. Epub 2009 Aug 20. PMID 19696119
- [Background] Cook G, Burton L, Hoogenboom BJ, Voight M. Functional movement screening: the use of fundamental movements as an assessment of function-part 2. Int J Sports Phys Ther. 2014 Aug;9(4):549-63. PMID 25133083